CLINICAL TRIAL: NCT05457361
Title: Venetoclax Combined With Azacitidine Plus Homoharringtonine Versus Venetoclax Combined With Azacitidine for Relapsed/Refractory Acute Myeloid Leukemia：an Open-label, Multicentre, Randomised Phase 3 Trial
Brief Title: VAH Versus VA for Salvage Therapy of R/R-AML
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Shenzhen Hospital of Southern Medical University (Other); Peking University Shenzhen Hospital (Other); Shenzhen Second People's Hospital (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Southern Medical University, China (Other); First People's Hospital of Chenzhou (Other); The Affiliated Hospital of Qingdao University (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Department director, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAH vs VA-2022
Record Dates: First submitted 2022-03-08; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Venetoclax Combined With Azacitidine Plus Homoharringtonine; Venetoclax Combined With Azacitidine
Keywords: Relapsed/refractory acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAH regimen (Experimental): VEN begins at 100 mg on day 1 and increases stepwise over 3 days to reach the target dose of 400 mg (100 mg, 200 mg, 400 mg); dosing is continued at 400 mg per day from day 4 through day 14; azacitidine (75 mg/m²) is administered subcutaneously on days 1-7, and HHT (1 mg/m²) on days 1-7.
  Interventions: Drug: VEN combined with azacitidine plus homoharringtonine
- VA regimen (Active Comparator): The use of VEN is just the same as it dose in VAH regimen except lasting for 28 days. The use of azacitidine is exactly the same as VAH group does.
  Interventions: Drug: VEN combined with azacitidine

INTERVENTIONS:
Drug: VEN combined with azacitidine plus homoharringtonine — VEN begins at 100 mg on day 1 and increases stepwise over 3 days to reach the target dose of 400 mg (100 mg, 200 mg, 400 mg); dosing is continued at 400 mg per day from day 4 through day 14; azacitidine (75 mg/m²) is administered subcutaneously on days 1-7, and HHT (1 mg/m²) on days 1-7.
  Arms: VAH regimen
Drug: VEN combined with azacitidine — The use of VEN is just the same as it dose in VAH regimen except lasting for 28 days. The use of azacitidine is exactly the same as VAH group does.
  Arms: VA regimen

SUMMARY:
This is a prospective, multi-center, phase 3 randomized controlled clinical study comparing VAH and VA regimens for the salvage treatment of the patients with relapsed/refractory AML. Approximately 164 subjects will be randomized in a 1:1 ratio to receive VAH regimen (82 subjects) or VA regimen (82 subjects) for salvage therapy. Randomization is done with permuted blocks (block size four), and implemented through an interactive web-based response system.

VAH regimen: VEN begins at 100 mg on day 1 and increases stepwise over 3 days to reach the target dose of 400 mg (100 mg, 200 mg, 400 mg); dosing is continued at 400 mg per day from day 4 through day 14; azacitidine (75 mg/m²) is administered subcutaneously on days 1-7, and HHT (1 mg/m²) on days 1-7.

VA regimen: The use of VEN is just the same as it dose in VAH regimen except lasting for 28 days. The use of azacitidine is exactly the same as VAH group does.

The primary endpoint was overall response rate (ORR) after 2 cycles of trial therapy.

The secondary endpoints were CRc after 2 cycles of trial therapy, overall survival (OS), event-free survival (EFS) and relapse at 2 year, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed/refractory AML The diagnosis of AML or relapsed AML was based on the criteria from NCCN, defined as recurrence of blasts in the peripheral blood (PB) or bone marrow (BM) blasts > 5% or development of extramedullary disease of patients after achieving a CR. Refractory AML was defined as no composite complete remission (CRc) and a reduction in bone marrow blasts of less than 50% after one cycle or no CRc after two cycles.
2. Age 18 to 65 years old with Eastern Cooperative Oncology Group (ECOG) performance status 0-2
3. Sign informed consent form, have the ability to comply with study and follow-up procedures

Exclusion Criteria:

1. Acute promyelocytic leukemia (AML subtype M3)
2. Previous exposure to the treatment of VEN-based regimen
3. Life expectancy less than 30 days after salvage therapy
4. Cardiac dysfunction (particularly congestive heart failure, unstable coronary artery disease and serious cardiac ventricular arrhythmias requiring antiarrhythmic therapy)
5. Respiratory failure ( PaO2 ≤60mmHg)
6. Hepatic abnormalities (total bilirubin ≥2 times the upper limit of normal [ULN], alanine aminotransferase or aspartate aminotransferase ≥2 times the ULN)
7. Renal dysfunction (creatinine ≥2 times the ULN or creatinine clearance rate < 30 mL/min)
8. ECOG performance status 3, 4 or 5
9. With any conditions not suitable for the trial (investigators' decision)
10. Active acute or chronic graft-versus-host disease (GVHD). Active acute GVHD or chronic GVHD was defined as GVHD requiring either at least 1 mg/kg per day of prednisone (or equivalent) or treatment beyond systemic corticosteroids.
11. Patients with pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | At the end of Cycle 2 (each cycle is 28 days)
  Overall response including CR/CRi and PR

SECONDARY OUTCOMES:
Composite complete remission rate | At the end of Cycle 2 (each cycle is 28 days)
  Composite complete remission including CR/CRi
Overall survival | From date of randomization until date of death from any cause, assessed up to 12 months.
  The time from enrolling to death or the last follow up
Event-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  The time from enrolling to no response, relapse, death or the last follow up
Relapse | 1 year
  The event of relapse
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Baseline to 30 day post the salvage therapy
  Haematological toxicity and non-haematological toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Department of Hematology,Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes